CLINICAL TRIAL: NCT04460274
Title: Time Series Model For Forecasting the Number of Covid-19 Cases Worldwide - A Prospective Cohort Study
Brief Title: Forecast Number of Covid-19 Cases Worldwide
Acronym: Covid19TmeSer
Status: Completed | Type: Observational
Sponsor: Turkish Ministry of Health Izmir Teaching Hospital (Other Government)
Responsible Party: Principal Investigator, Serhat Akay, Principal Investigator, Turkish Ministry of Health Izmir Teaching Hospital
Other Study IDs: TurkishMOHITH-TimeSeries
Record Dates: First submitted 2020-07-03; First posted 2020-07-07 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Covid-19
Keywords: Covid19, forecasting
MeSH Terms: conditions — COVID-19 | interventions — Boosting Machine Learning Algorithms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Model Building: Number of Covid-19 cases from December 31, 2019 to June 1, 2020 were used to build ARIMA model using Hyndman-Khandakar algorithm.
  Interventions: Other: Model Building
- Model Validation: Number of Covid-19 cases from June 2, 2020 to June 15, 2020 were used to forecast cases using the ARIMA model
  Interventions: Other: Model validation

INTERVENTIONS:
Other: Model Building — Model building
  Groups: Model Building
Other: Model validation — Model validation
  Groups: Model Validation

SUMMARY:
Coronavirus disease-19 (Covid-19) had an unprecedented effect on both nations and health systems. Time series modeling using Auto-Regressive Integrated Moving Averages (ARIMA) models have been used to forecast variables extensively mainly in statistics and econometrics. The investigators aimed to predict the total number of cases for Covid-19 using ARIMA models of time-series analysis.

DETAILED DESCRIPTION:
Coronavirus Disease 19 (Covid-19) is an infectious disease initially defined in December 2019 before becoming pandemic. Respiratory disease is the main form of disease causing acute respiratory distress as the main cause of death.

Increased number of cases worldwide had put an enormous load on public health resulting lockdowns, quarantines and curfews. Predicting number of cases is hard as the increment of cases between communities differ.

Time series had been used in different fields of science to predict, such as signal processing, mathematical finance, weather prediction. In medicine, time series analysis were used in number of admitted patients to hospitals. Aim of this study is to predict the total number of Covid-19 cases worldwide using time series anaylsis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed case of Covid-19

Exclusion Criteria:

* Cases not reported

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population consists all confirmed cases of Covid-19 reported from Situation Dashboard of the European Center for Disease Prevention and Control website Coronavirus 19 Situation Report
Sampling Method: Non-Probability Sample
Enrollment: 7882471 (Actual)
Dates: Start 2019-12-31 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Number of Confirmed cases of Covid-19 | December 31, 2019 to June 15, 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Republic of Turkey, Health Sciences University, Izmir Bozyaka Education and Training Hospital, Izmir, Turkey (Türkiye)